CLINICAL TRIAL: NCT03529227
Title: Prospective One-center Open Label Observational Efficacy & Safety Study of Chlorambucil & Obinutuzumab in Treatment of Unfit Patients With Untreated Chronic Lympho Leukemia With Comorbidities
Brief Title: Gazyva Infusion Reaction Investigation
Acronym: GAIRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Healthy Future (Other)
Responsible Party: Sponsor
Other Study IDs: ML40194
Record Dates: First submitted 2018-03-29; First posted 2018-05-18 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chlorambucil; obinutuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study evaluate safety and effectiveness of chlorambucil and obinutuzumab in routine clinical practice in patients with chronic lymphatic leukemia and with certain comorbidities (any cardiac pathology, diabetes mellitus (DM), kidney pathology or cytopenia), whom obinutuzumab & chlorambucil have been applied according to indications before enrollment in the study.

DETAILED DESCRIPTION:
MRD (Minimal residual disease) evaluation was chosen as a primary measure outcome as it is considered as prognostic marker for long-term progression freee survival (PFS) and as a potential therapeutic goal in chronic lymphocytic leukemia/ CLL .

Minimal residual disease (MRD-negative) is assessed in the clinic by 8-color flow cytometry giving the sensitivity level of MRD detection 10-5; MRD is measured in real clinical practice at this clinical center according to National recommendations in diagnostics and treatment of lymphoproliferative disorders.

To achieve study objectives medical patients' charts will be analyzed retrospectively. In the frame of this program 104 patients' charts treated in defined clinical site, are planned to be analyzed. This number of patients corresponds to the patient flow with this pathology at a defined clinical site for 1 years.

Data collection is considered to be retrospective as data will be transferred to e-CRF from patient medical charts. During this study no further specific extra procedures for data gathering is expected.

But since patients included in the study will be at the center of ongoing therapy, the study was called a prospective.

ELIGIBILITY:
Inclusion Criteria:

1. CD20+/ (cluster of differentiation antigen 20 positive) B-CLL pts on the 1st line treatment therapy, whom have been already applied Obinutuzumab and chlorambucil
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group Scale (ECOG) 0-2.
4. Total Chronic Illness Resources Survey scale (CIRS) score >6 or creatinine clearance <70 ml/min or both for patients ≥ 18 years old or all CLL pts ≥ 75 years old
5. Any cardiac pathology/ diabetes mellitus/ kidney pathology/ cytopenia (Hb <100 g/l, Platelets < 100 x 109/l)
6. Life expectancy more than 6 months according to the physician's opinion.
7. Signed informed consent that allow personal data and data that refer to patient confidentiality processing

Exclusion Criteria:

The refusal of the patient to participate in the observational study and the withdrawal of informed consent that allow processing of personal data and data that refer to patient confidentiality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected to include 104 patient with primary diagnosed CLL elder 18 years with certain comorbidities as any cardiac pathology/ diabetes mellitus/ kidney pathology/ cytopenia (Hb <100 g/l, Platelets < 100 x 109/l) after Obinutuzumab + chlorambucil are applied as the 1st line treatment .
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2018-03-31 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
MRD status of CLL patients with comorbidities | 3 months after the last dose of study treatment
  Number of patients with positive and negative MRD status

SECONDARY OUTCOMES:
Response Rate (ORR) | 3 months after last dose administration
  Frequency of the overall response in patients with CLL using the Chlorambucil + Obinutuzumab (G-Clb) therapy regimen (N,%)
Progression free survival (PFS) by the Kaplan-Meier method | 3 months after last dose administration
  Time to full remission in patients with CLL using Chlorambucil + Obinutuzumab (G-Clb) therapy regimen (month) calculated by the Kaplan-Meier method
Duration of response (DOR) by the Kaplan-Meier method | 3 months after last dose administration
  Time to partial remission in patients with CLL using Chlorambucil + Obinutuzumab (G-Clb) therapy regimen (month) calculated by the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Eugeny A Nikitin, MD, Principal Investigator — "The State Budgetary Moscow Healthcare Institution Clinical Hospital named after S.P. Botkin of Moscow Health Department"
Locations (2):
- Russia (2):
  - The State Budgetary Moscow Healthcare Institution Clinical Hospital named after S.P. Botkin of Moscow Health Department"., Moscow
  - The State Budgetary Moscow Healthcare Institution Clinical Hospital named after S.P. Botkin of Moscow Health Department, Moscow

REFERENCES:
- [Result] Под ред. А.Д. Каприна, В.В. Старинского, Г.В. Петровой, "Злокачественные новообразования в России в 2015 году (заболеваемость и смертность)" - М.: МНИОИ им. П.А. Герцена - филиал ФГБУ "НМИРЦ" Минздрава России - 2017. - ил. - 250 с. ISBN 978-5-85502-227-8.
- [Result] Российские клинические рекомендации по диагностике и лечению лимфопролиферативных заболеваний. Под руководством профессора И.В. Поддубной, профессора В.Г. Савченко. М., 2016. - 412 с.
- [Result] Kwok M, Rawstron AC, Varghese A, Evans PA, O'Connor SJ, Doughty C, Newton DJ, Moreton P, Hillmen P. Minimal residual disease is an independent predictor for 10-year survival in CLL. Blood. 2016 Dec 15;128(24):2770-2773. doi: 10.1182/blood-2016-05-714162. Epub 2016 Oct 3. PMID 27697770